CLINICAL TRIAL: NCT03135340
Title: Comparison of Wide-Awake Local Anesthesia vs. Regional/General Anesthesia for Hand Flexor Tendon Repair in Zones I and II: a Prospective Randomized Controlled Trial
Brief Title: Wide-Awake Local Anesthesia vs. Regional/General Anesthesia for Flexor Tendon Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Organization: Western University, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UWO7788705772
Record Dates: First submitted 2016-12-06; First posted 2017-05-01 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-04

CONDITIONS: Tendon Injury - Hand
MeSH Terms: interventions — Anesthesia, Conduction

STUDY DESIGN:
Intervention Model Description: Two groups. One interventional group and one control group with random allocation as described below.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to the treatment received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WALANT (Experimental): These patients will receive local anesthetic for flexor tendon repair injected directly into the operative site on the hand. The local anesthetic used 1% lidocaine with 1:100,000 epinephrine.
  Interventions: Procedure: WALANT; Drug: WALANT Injection
- General/regional anesthesia (Active Comparator): These patients will receive general/regional anesthesia for flexor tendon repair. This is ropivacaine 0.5% injected by an anesthetist under image-guidance in the axillary region of the arm. If the regional anesthesia is not functioning at the time of OR, this is converted to a general anesthetic as per standard protocol.
  Interventions: Procedure: General/regional anesthesia; Drug: Regional Anesthetic Injection

INTERVENTIONS:
Procedure: WALANT — These patients will receive local anesthetic for flexor tendon repair injected directly into the operative site on the hand. The local anesthetic used 1% lidocaine with 1:100,000 epinephrine.
  Arms: WALANT
Procedure: General/regional anesthesia — These patients will receive general/regional anesthesia for flexor tendon repair. This is ropivacaine 0.5% injected by an anesthetist under image-guidance in the axillary region of the arm. If the regional anesthesia is not functioning at the time of OR, this is converted to a general anesthetic as per standard protocol.
  Arms: General/regional anesthesia
Drug: WALANT Injection — 1% lidocaine with 1:100,000 epinephrine injected directly into operative site. The typical quantity is 5-10cc aliquots.
  Arms: WALANT
Drug: Regional Anesthetic Injection — 0.5% ropivacaine injected under ultrasound guidance into the axilla. The typical quantity is 30-40cc aliquots.
  Arms: General/regional anesthesia

SUMMARY:
Wide-awake hand surgery with local anesthetic, no tourniquet and no sedation (WALANT) is increasingly utilized. Conventional anesthesia for hand surgery involves a patient with a block, unable to perform motor function in the arm, and with patient either intubated or sedated, unable to follow surgeon instructions intra-operatively. Flexor tendon repair with a wide awake and cooperative patient is routinely performed successfully at some centres. This method provides several potential benefits including being able to have the patient actively flex the digit and visualize the repair site to assess for any tendon gapping at the repair site, ensure adequate approximation, gliding and absence of triggering. There have not been any prospectively collected randomized controlled trials comparing wide awake vs. regional/general anesthesia in flexor tendon repair. The purpose of our study is to assess for differences in early outcomes including stiffness, patient satisfaction and early complications in wide-awake anesthesia when compared to general/regional anesthesia for flexor tendon repair in zones I and II. Our hypothesis is that there is a lower complication rate and better outcomes when using wide-awake flexor tendon repair.

DETAILED DESCRIPTION:
Primary repair for flexor tendon lacerations remain the standard of care. However, despite recent advances in knowledge of tendon healing, suture material, and post-operative protocols, outcomes have been reported as fair or poor in 7-20% of patients. Complications encountered include adhesion formation, development of joint contractures, tendon rupture, triggering, bowstringing and quadrigia.

Wide-awake flexor tendon repair using local anesthesia and epinephrine with no tourniquet has been described. Safety of epinephrine in digits makes it possible, and epinephrine-induced vasoconstriction precludes the need for a tourniquet and cautery.This approach allows a wide-awake, comfortable, non-sedated, cooperative, tourniquet-free patient to test the freshly repaired tendon with full active range of motion intraoperatively. The surgeon can inspect for bunching, gapping, and triggering of the repair site in an active fashion. Thus, an opportunity is available to revise the repair, trim or add extra sutures, revise pulley reconstruction, or de-bulk tendons before wound closure. This could mean that a higher quality repair is possible and could guide post-operative rehabilitation. It follows that if the patient is unable to achieve total active range of motion intraoperatively they will not be able to postoperatively and may end up requiring a tenolysis. Lalonde and colleagues looked retrospectively at their 15 years of experience using WALANT with the hypothesis that this technique decreased their post-operative rupture rate. With 122 patients there were only 3 ruptures, all due to unexpected forceful movements. Contraindications of this technique include patients who are unable or unwilling to tolerate an operation while awake, pediatric patients, those who are mentally impaired, and complex trauma.

Improved compliance with postoperative therapy is also reported after patients visualize the repair in real time and gain a better understanding of limitations and expectations. Patient buy-in to the rehabilitation process is potentially improved if the surgeon can use the operative time to educate the patient, show them the repair, and manage expectations since the patient is wide-awake and coherent. Wide-awake flexor tendon repair could also improve surgeon confidence in initiating a true active motion therapy protocol when the surgeon visualizes the absence of gapping with full finger flexion. Initiation of early active motion could subsequently improve ultimate post-operative range of motion and patient satisfaction. The advent of wide-awake flexor tendon repair could have economic implications as well given that fewer resources are theoretically used for the procedure.

Currently there are no prospective randomized controlled studies evaluating outcomes in flexor tendon repairs that have utilized a wide-awake anaesthesia protocol and comparing outcomes with traditional repair techniques.

The purpose of this study is to evaluate and compare outcomes of WALANT (wide-awake, local anesthetic, no tourniquet) when compared to traditional general/regional anesthetic for flexor tendon repairs in zone I and II.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* acute single or multiple digit complete flexor tendon lacerations in zones I or II presenting to attending physicians who agree to participate in the study.

Exclusion Criteria:

* gross wound contamination
* segmental tendon loss
* associated finger fractures
* sub-acute or chronic ruptures (ruptures > 6 weeks old)
* active or previous infection in the wound bed
* requirement of delayed repair
* complex or multisystem injuries
* multiple digit injuries
* significant joint injuries
* amputations (replants)
* mangled hand injuries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2033-11 (Estimated)

PRIMARY OUTCOMES:
Complication rate | 1 year
  Infection requiring antibiotics, tendon rupture, stiffness or contracture requiring tenolysis

SECONDARY OUTCOMES:
Total active range of motion | 1 year
  This is measured as active digit motion measured at the proximal interphalangeal and distal interphalangeal joints with use of a goniometer by a hand therapist
Strickland Criteria Score | 1 year
  The sum of active ranges of motion of the proximal interphalangeal (PIP) and distal interphalangeal (DIP) joints. Then the percentage is calculated, in comparison to the contralateral side. The scores are then recorded as one of four categories: Excellent: 85-100%, Good: 70-84%, Fair: 50-69, Poor: 0-49%
Pain of procedure by visual analogue scale (VAS) | 1 week
  Measured on visual analogue scale on a 10cm line and scored out of 10 (0 being no pain and 10 being maximum pain)
Pain of procedure by pain diary | 1 week
  The pain diary is used by the patient at home to record subjective daily pain from 0-10 at a predetermined time every day.
Subjective anxiety | 1 week
  anxiety surrounding procedure as measured on a VAS (from 0 being no anxiety to 10 being maximum anxiety)
Repeat procedure question | 1 week
  The patient is asked whether or not they would undergo the procedure the same way again (yes or no).
DASH (disabilities of the arm, shoulder and hand) Score | 1 year
  This outcome instrument is a thirty-question self-reported survey of function and symptoms in patients with upper extremity disorders. Scores range from 0 (no disability) to 100 (completely disabled).

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Grewal, MD MSc FRCSC, Principal Investigator — Western University, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verdan CE. Half a century of flexor-tendon surgery. Current status and changing philosophies. J Bone Joint Surg Am. 1972 Apr;54(3):472-91. No abstract available. PMID 4560071
- [Background] Saldana MJ, Chow JA, Gerbino P 2nd, Westerbeck P, Schacherer TG. Further experience in rehabilitation of zone II flexor tendon repair with dynamic traction splinting. Plast Reconstr Surg. 1991 Mar;87(3):543-6. doi: 10.1097/00006534-199103000-00023. PMID 1998024
- [Background] Lilly SI, Messer TM. Complications after treatment of flexor tendon injuries. J Am Acad Orthop Surg. 2006 Jul;14(7):387-96. doi: 10.5435/00124635-200607000-00001. PMID 16822886
- [Background] Wilhelmi BJ, Blackwell SJ, Miller J, Mancoll JS, Phillips LG. Epinephrine in digital blocks: revisited. Ann Plast Surg. 1998 Oct;41(4):410-4. doi: 10.1097/00000637-199810000-00010. PMID 9788222
- [Background] Denkler K. A comprehensive review of epinephrine in the finger: to do or not to do. Plast Reconstr Surg. 2001 Jul;108(1):114-24. doi: 10.1097/00006534-200107000-00017. PMID 11420511
- [Background] Nodwell T, Lalonde D. How long does it take phentolamine to reverse adrenaline-induced vasoconstriction in the finger and hand? A prospective, randomized, blinded study: The Dalhousie project experimental phase. Can J Plast Surg. 2003 Winter;11(4):187-90. doi: 10.1177/229255030301100408. PMID 24009436
- [Background] Higgins A, Lalonde DH, Bell M, McKee D, Lalonde JF. Avoiding flexor tendon repair rupture with intraoperative total active movement examination. Plast Reconstr Surg. 2010 Sep;126(3):941-945. doi: 10.1097/PRS.0b013e3181e60489. PMID 20463621
- [Background] Lalonde DH. Wide-awake flexor tendon repair. Plast Reconstr Surg. 2009 Feb;123(2):623-625. doi: 10.1097/PRS.0b013e318195664c. No abstract available. PMID 19182622
- [Background] Lalonde DH. An evidence-based approach to flexor tendon laceration repair. Plast Reconstr Surg. 2011 Feb;127(2):885-890. doi: 10.1097/PRS.0b013e31820467b6. PMID 21285792
- [Background] Momeni A, Grauel E, Chang J. Complications after flexor tendon injuries. Hand Clin. 2010 May;26(2):179-89. doi: 10.1016/j.hcl.2009.11.004. PMID 20494744
- [Background] Dowd MB, Figus A, Harris SB, Southgate CM, Foster AJ, Elliot D. The results of immediate re-repair of zone 1 and 2 primary flexor tendon repairs which rupture. J Hand Surg Br. 2006 Oct;31(5):507-13. doi: 10.1016/j.jhsb.2006.06.006. Epub 2006 Aug 22. PMID 16930791
- [Background] Mustoe TA, Buck DW 2nd, Lalonde DH. The safe management of anesthesia, sedation, and pain in plastic surgery. Plast Reconstr Surg. 2010 Oct;126(4):165e-176e. doi: 10.1097/PRS.0b013e3181ebe5e9. PMID 20885206
- [Background] Strickland JW. Results of flexor tendon surgery in zone II. Hand Clin. 1985 Feb;1(1):167-79. PMID 4093459